CLINICAL TRIAL: NCT02611297
Title: Cryoprobe Transbronchial Lung Biospy in Patients With Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Germans Trias i Pujol Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIBSP-CRI-2013-142
Record Dates: First submitted 2015-05-21; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Lung Diseases; Interstitial Disease
Keywords: Cryoprobes; Cryobiopsy; Transbronchial lung biopsy
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transbronchial lung biopsy with cryoprobe (Other)
  Interventions: Procedure: Cryoprobe

INTERVENTIONS:
Procedure: Cryoprobe

SUMMARY:
The purpose of this study is to evaluate the the diagnostic yield and safety of transbronchial lung biopsies (TBLB) with cryoprobe in patients with mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Patients with mechanical ventilation.
* Patients with diffuse lung disease of unknown etiology.
* Need for confirming/excluding a diagnosis, with therapeutical and prognosis implications.
* Inform consent signed by family.

Exclusion Criteria:

* Use of anticoagulant therapy or presence of a coagulation disorder (abnormal platelets counts, international normalized ratio > 1.5).
* Comorbidities that could increase the risk of the TBLB.
* Bullous emphysema.
* Hemoptysis, pneumothorax.
* Severe respiratory insufficiency requiring PEEP >12 cm H2O

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2013-11; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events related to transbronchial lung biopsy (TBLB) with cryoprobe | 27 months

SECONDARY OUTCOMES:
Diagnostic yield of transbronchial lung biopsy (TBLB) obtained by cryoprobes | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Pajares, MD, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (3):
- Spain (3):
  - Germans Tries i Pujol Hospital, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Clinic de Barcelona, Barcelona, Barcelona